CLINICAL TRIAL: NCT07329452
Title: Menu to Meal (M2M): Evaluating the Effectiveness of a Digital Nutritional Labeling Intervention in Hispanic Restaurant Settings
Brief Title: Menu to Meal (M2M) Menu Labeling Intervention Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Hyunjung Lee, Assistant Professor, Texas A&M University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY2025-1204
Record Dates: First submitted 2025-11-24; First posted 2026-01-09 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Behavior, Eating
Keywords: nutrition labeling; menu labeling; Augmented reality (AR); Artificial intelligence (AI); Dietary behavior; Hispanic population; Chronic disease prevention; Obesity; Type 2 diabetes; Cardiovascular disease; Calorie intake; Sodium intake; Saturated fat; Food choice; Health disparities; Behavioral intervention; Digital health intervention; Restaurant nutrition; Health literacy; Theory of Planned Behavior (TPB); Social Cognitive Theory (SCT); Behavioral Nutrition
MeSH Terms: conditions — Feeding Behavior; Obesity; Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This study uses a within-site, quasi-experimental design at two independently owned Hispanic restaurants. The intervention consists of three sequential conditions: (1) a baseline phase with the standard menu, (2) a paper menu phase featuring bilingual nutrition labels, and (3) a digital menu phase using a mobile app enhanced with augmented reality (AR) and artificial intelligence (AI) technologies. Each condition enrolls distinct participants to compare the effects of different menu labeling formats on ordering behavior and psychosocial outcomes. The restaurants serve as their own controls, allowing for direct comparison of menu formats within the same real-world setting.
Masking Description: Participants in this study will be partially blinded to the specific aims of the intervention to minimize bias. While they will be aware they are participating in a study about menu use and food choices, they will not be informed of the detailed differences or hypotheses related to the nutrition labeling formats to reduce influence on their ordering behavior. Research staff collecting data will also be trained to maintain neutrality, but full masking is not possible due to the visible differences in menu formats across study phases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline condition (No Intervention): Standard menu with no nutrition information.
- Paper menu condition (Active Comparator): Bilingual paper menus display numeric and icon-based nutrition information, including calories, saturated fat, and sodium.
  Interventions: Behavioral: Paper menu
- AR/AI digital menu condition (Experimental): Mobile app providing interactive nutrition information and personalized guidance based on dietary preferences.
  Interventions: Behavioral: Digital menu condition

INTERVENTIONS:
Behavioral: Paper menu — Paper menu with bilingual nutrition labels
  Arms: Paper menu condition
Behavioral: Digital menu condition — AR/AI-enhanced digital menu giving interactive nutrition guidance
  Arms: AR/AI digital menu condition

SUMMARY:
This study evaluates the impact of culturally tailored menu labeling interventions on psychosocial factors and ordering behavior among customers in two independently owned Hispanic restaurants in East-Central Texas. Participants will be exposed to one of three sequential menu conditions at each restaurant: (1) a standard menu without nutrition information, (2) a paper menu with bilingual nutrition labels, or (3) a digital menu app enhanced with Augmented Reality (AR) and Artificial Intelligence (AI) providing interactive nutrition guidance. The study will assess whether menu formats influence nutrition literacy, decision-making confidence, self-efficacy, attitudes, behavioral intentions, and actual ordering behavior. Data will be collected through surveys, purchase receipts, and app interaction logs.

DETAILED DESCRIPTION:
Detailed Description:

This study aims to design and evaluate a culturally tailored, bilingual menu labeling intervention incorporating AR and AI features in small, independently owned Hispanic restaurants. The intervention seeks to promote informed food ordering by targeting psychosocial constructs known to influence food choice. Three sequential conditions will be implemented: (1) baseline with standard menus and no nutrition labels, (2) paper menus with visible bilingual nutrition labels, and (3) a digital AR/AI-enhanced menu.

Guided by the Theory of Planned Behavior and Social Cognitive Theory, the study focuses on constructs such as decision-making confidence, self-efficacy, subjective norms, and perceived behavioral control. The two primary objectives are to (1) develop a culturally informed digital menu labeling tool and (2) evaluate its effectiveness compared with standard and paper menu formats in shaping psychosocial factors and actual ordering behavior.

Participants will be recruited during restaurant visits and exposed to the menu condition corresponding to their visit timing. Surveys will be administered before ordering to assess psychosocial factors, label awareness, and behavioral intentions. A formative needs assessment conducted prior to implementation will ensure cultural and linguistic appropriateness. Findings will provide evidence on the effectiveness of innovative, theory-informed digital interventions in promoting informed food choices in culturally specific restaurant settings not subject to federal nutrition labeling requirements.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Patrons dining at participating Hispanic restaurants during designated study hours
* Able to read and speak English or Spanish
* Willing and able to provide informed consent
* Pregnant women are eligible to participate, as the study procedures pose minimal risk

Exclusion Criteria:

* Minors under 18 years of age
* Individuals with visual or cognitive impairments that prevent interaction with the menu formats or AR/AI technology
* Individuals who have participated in a prior phase of the study
* Restaurant staff involved in study implementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Attitudes Toward Healthy Menu Choices | Immediately after the intervention (menu exposure)
  Attitudes toward selecting healthier menu items, assessed using a study-developed questionnaire informed by the Theory of Planned Behavior. The questionnaire consists of agreement-scale items evaluating whether choosing healthier foods is important, beneficial, and enjoyable.
  Measurement Tool:
  Study-developed Attitudes Toward Healthy Menu Choices Questionnaire (5-point agreement Likert scale)
  Scale Description and Coding:
  1. = Strongly disagree
  2. = Disagree
  3. = Neither agree nor disagree
  4. = Agree
  5. = Strongly agree
  Unit of Measure:
  Mean attitude score (range: 1 to 5)
  Scale Range and Direction:
  Scores range from 1 to 5. Higher scores indicate more positive attitudes toward choosing healthier menu items.
Intention to Make Healthier Food Choices | Immediately after the intervention (menu exposure)
  Intention to choose healthier menu items, assessed using a study-developed questionnaire informed by the Theory of Planned Behavior.
  Measurement Tool:
  Study-developed Healthy Eating Intention Questionnaire (5-point agreement Likert scale)
  Scale Description and Coding:
  1. = Strongly disagree
  2. = Disagree
  3. = Neither agree nor disagree
  4. = Agree
  5. = Strongly agree
  Unit of Measure:
  Intention score (range: 1 to 5)
  Scale Range and Direction:
  Scores range from 1 to 5. Higher scores indicate stronger intention to choose healthier menu items.
Perceived Behavioral Control Over Healthy Menu Choices | Immediately after the intervention (menu exposure)
  Perceived behavioral control over choosing healthier menu items, assessed using a study-developed questionnaire informed by the Theory of Planned Behavior.
  Measurement Tool:
  Study-developed Perceived Behavioral Control Questionnaire (5-point agreement Likert scale)
  Scale Description and Coding:
  1. = Strongly disagree
  2. = Disagree
  3. = Neither agree nor disagree
  4. = Agree
  5. = Strongly agree
  Unit of Measure:
  Perceived behavioral control score (range: 1 to 5)
  Scale Range and Direction:
  Scores range from 1 to 5. Higher scores indicate greater perceived control over choosing healthier menu items.
Self-Efficacy for Using Nutrition Information When Ordering | Immediately after the intervention (menu exposure)
  Self-efficacy for using nutrition information to guide food choices, assessed using a study-developed questionnaire informed by Social Cognitive Theory.
  Measurement Tool:
  Study-developed Nutrition Information Self-Efficacy Questionnaire (5-point agreement Likert scale)
  Scale Description and Coding:
  1. = Strongly disagree
  2. = Disagree
  3. = Neither agree nor disagree
  4. = Agree
  5. = Strongly agree
  Unit of Measure:
  Mean self-efficacy score (range: 1 to 5)
  Scale Range and Direction:
  Scores range from 1 to 5. Higher scores indicate greater confidence in using nutrition information to make food choices.
Awareness of Nutrition Information on the Menu | Immediately after the intervention (menu exposure)
  Awareness of nutrition information on the menu, assessed using a study-developed self-report item asking whether the participant noticed or looked at nutrition information while viewing the menu.
  Measurement Tool:
  Study-developed Awareness of Nutrition Information Item (binary response)
  Scale Description and Coding:
  0 = No, did not notice or look at nutrition information
  1 = Yes, noticed or looked at nutrition information
  Unit of Measure:
  Percentage of participants reporting awareness (response = 1)
  Scale Range and Direction:
  Values range from 0 to 1. A value of 1 indicates awareness of nutrition information.
  How the Percentage Is Derived:
  The percentage is calculated as the proportion of participants with a response of 1 (Yes) among all participants who completed the questionnaire.
Use of Nutrition Information to Inform Menu Selection | Immediately after the intervention (menu exposure)
  Use of nutrition information to inform menu selection, assessed using a study-developed self-report item asking the extent to which nutrition information influenced the participant's food choice.
  Measurement Tool:
  Study-developed Nutrition Information Influence Item (5-point Likert scale)
  Scale Description and Coding:
  1. = Not at all
  2. = A little
  3. = Somewhat
  4. = Mostly
  5. = Completely
  Unit of Measure:
  Percentage of participants reporting use of nutrition information, defined as responses of 4 or 5
  Scale Range and Direction:
  Scores range from 1 to 5. Higher values indicate greater influence of nutrition information on choice.
  How the Percentage Is Derived:
  The percentage is calculated as the proportion of participants with responses of 4 or 5 among all participants who completed the questionnaire.

SECONDARY OUTCOMES:
Total Energy Ordered per Customer Order | Immediately after the intervention (menu exposure)
  Total energy content of menu items ordered by each participant, calculated using receipt-based ordering data linked to laboratory-tested and standardized recipe-based nutrient analysis conducted as part of the Menu2Meal (M2M) intervention.
  Measurement Tool:
  Receipt-based nutrient calculation using laboratory-tested and standardized nutrient databases
  Unit of Measure:
  Mean kilocalories (kcal) per customer order
Saturated Fat Content of Menu Items Ordered | Immediately after the intervention (menu exposure)
  Total saturated fat content of menu items ordered by each participant, calculated by summing grams of saturated fat from all items ordered, using laboratory-tested and standardized recipe-based nutrient values.
  Measurement Tool:
  Receipt-based nutrient calculation using laboratory-tested and standardized nutrient databases
  Unit of Measure:
  Mean grams (g) of saturated fat per customer order
Sodium Content of Menu Items Ordered | Immediately after the intervention (menu exposure)
  Total sodium content of menu items ordered by each participant, calculated by summing milligrams of sodium from all items ordered, using laboratory-tested and standardized recipe-based nutrient values.
  Measurement Tool:
  Receipt-based nutrient calculation using laboratory-tested and standardized nutrient databases
  Unit of Measure:
  Mean milligrams (mg) of sodium per customer order
Dietary Fiber Content of Menu Items Ordered | Immediately after the intervention (menu exposure)
  Total dietary fiber content of menu items ordered by each participant, calculated by summing grams of dietary fiber from all items ordered, using laboratory-tested and standardized recipe-based nutrient values.
  Measurement Tool:
  Receipt-based nutrient calculation using laboratory-tested and standardized nutrient databases
  Unit of Measure:
  Mean grams (g) of dietary fiber per customer order
Added Sugar Content of Menu Items Ordered | Immediately after the intervention (menu exposure)
  Total added sugar content of menu items ordered by each participant, calculated by summing grams of added sugars from all items ordered, using laboratory-tested and standardized recipe-based nutrient values.
  Measurement Tool:
  Receipt-based nutrient calculation using laboratory-tested and standardized nutrient databases
  Unit of Measure:
  Mean grams (g) of added sugars per customer order

CONTACTS AND LOCATIONS:
Overall Officials: Hyunjung Lee, PhD, Principal Investigator — Department of Nutrition, Texas A&M University
Locations (1):
- Local Restaurant Site, Bryan, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in the publication will be shared, including baseline characteristics, outcome measures, and adverse event data. Data will be available beginning 6 months after publication for researchers who provide a methodologically sound proposal. Requests should be submitted to the corresponding author and will require a data use agreement in accordance with institutional and regulatory policies.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be made available beginning approximately 6 months after publication of the primary results and will remain available for 2 years.
Access Criteria: Researchers who wish to access the de-identified individual participant data (IPD) and supporting documents should submit a written request to the corresponding author. Requests must include a methodologically sound research proposal describing the intended analyses and purpose of data use. Access will be granted to qualified researchers upon approval of the proposal and execution of a data use agreement in accordance with Texas A&M University and applicable regulatory requirements. Data will be transferred using a secure institutional data-sharing platform.